CLINICAL TRIAL: NCT01375881
Title: Post Authorization Non-interventional Study in HIV1-Infected Patients Starting or Already in Treatment With Darunavir
Brief Title: Non-interventional Study on Use of Darunavir With Ritonavir in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag S.p.A. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017641; TMC114HIV4042 (Other: Janssen-Cilag S.p.A., Italy)
Record Dates: First submitted 2011-06-09; First posted 2011-06-17 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: HIV Infections
Keywords: HIV; darunavir; ritonavir; Prezista; naive; experienced
MeSH Terms: conditions — HIV Infections | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Observational Model: Cohort

GROUPS / COHORTS (1):
- 001: darunavir/ritonavir plus background regimen darunavir/ritonavir oral use in naive and experienced patients at approved dosages
  Interventions: Drug: darunavir/ritonavir plus background regimen

INTERVENTIONS:
Drug: darunavir/ritonavir plus background regimen — darunavir/ritonavir, oral use, in naive and experienced patients at approved dosages

SUMMARY:
The purpose of this non-interventional study is a description of use of darunavir in daily practice, in retrospective and perspective manner. Darunavir will be prescribed in the usual manner and in accordance with the terms of marketing authorization. The assignment of a patient to a particular therapeutic strategy will not be decided in advance by this study protocol but instead, it will be part of the current clinical practice. The prescription of the medicinal product will be clearly separated from the decision to include the patient in the study. No additional diagnostic or monitoring procedures will be applied to the patients, and epidemiological methods will be used for the analysis of collected data. After having agreed with the patient on starting treatment with darunavir, and provided that all inclusion and exclusion criteria apply, the physician will document the patient's data. Patients will be observed for at least 48 weeks from baseline visit except for those who withdraw from the study earlier. Patients data will be collected at approximately 0, 1, 3 and 6 months after starting treatment and subsequently every 3 months in accordance with routine practice. The expected number of patients to enroll is about 900. The patients will be treated with darunavir according to the Italian label. The patient must be withdrawn from the study if the treatment with darunavir has been stopped. A last evaluation must be documented when possible, and a resistance test will be collected if available for patients discontinuing for virologic failure. At the end of study visit, information on therapy given after darunavir discontinuation will be collected. For patients discontinuing for virologic failure, data will be collected until the end of the present study, and at least two consecutive measurements of viral load after starting new antiretroviral therapy will be collected, if available. All data collected must be the result of the normal medical care of the patient. The patient's baseline data will be collected within the first week before darunavir administration (at Visit 1). For patients already in treatment with darunavir, baseline and follow up data will be collected retrospectively and prospectively. Further data collection will occur approximately at 1, 3, and 6 months and subsequently about every 3 months according to routine practice, after initiating darunavir treatment.

DETAILED DESCRIPTION:
The patient's baseline data will be collected within the first week before darunavir administration, Visit 1. For patients already in treatment with darunavir, outside the Early Access Program, baseline and follow-up data will be collected retrospectively and prospectively. For patients switched to commercial darunavir from the Early Access Program and already in treatment with darunavir, Baseline Visit data will be collected from the Early Access Program Baseline Visit. For patients already in treatment with darunavir outside the Early Access Program, baseline data will be collected retrospectively starting from the first darunavir intake. For all patients, laboratory examination results collected within 6 months before darunavir treatment starts will be considered as baseline data. For patients switched to commercial darunavir from the Early Access Program and already in treatment with darunavir, Visit 2 won't be performed. For patients starting commercial darunavir or already in treatment with commercial darunavir outside the Early Access Program, laboratory exams related to follow-up visits, Visit 2 onward, can be performed within a time window of one month before or after the corresponding visit date. Further data collection will occur approximately at 1, 3, and 6 months and subsequently about every 3 months according to routine practice, after initiating darunavir treatment. If a patient stops treatment with darunavir at any time, the end of study visit should be performed as soon as possible. Darunavir film-coated tablet, orally administered. Orange, oval-shaped tablet, debossed with 400MG or 600MG or 300MG on one side and TMC on the other side. Duration of observation minimum 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Eligible for inclusion in this non-interventional study are adult patients in need of treatment with darunavir according to Italian label or already in treatment

* Having provided a signed and dated Informed Consent Form

Exclusion Criteria:

* A known hypersensitivity to darunavir or to any of its excipients
* Severe hepatic impairment described as Child-Pugh class C
* Pregnancy or lactation
* Patient previously treated with darunavir that was discontinued for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient using darunavir and ritonavir in clinical practice according to label in Italy. Both naive and experienced patients are allowed to enter the study
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Measurement of viral load, as an assessment of efficacy | At least 48 weeks

SECONDARY OUTCOMES:
Immunological response, as measured by CD4 cells count | At least 48 weeks
Impact on Health-related Quality of Life after switching to a darunavir containing regimen in accordance to the approved indication | At least 48 weeks
Neuropsychological impairment at baseline and after switching to a darunavir containing regimen in accordance to the approved indication | At least 48 weeks
Assessments of non-categorized information gathered about treatment switch to and from darunavir | At least 48 weeks
Number of patients with adverse events, as a measure of safety | At least 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag S.p.A. Clinical Trial, Study Director — Janssen-Cilag S.p.A.